CLINICAL TRIAL: NCT07380828
Title: Multicenter Observational Prospective Study of Cardio-reno- Hepato -Metabolic Disease in Chronic Heart Failure
Brief Title: CArdio-Reno- Hepato -MEtabolic Disease iN Chronic Heart Failure (CARMEN-CHF)
Acronym: CARMEN-CHF
Status: Not yet recruiting | Type: Observational
Sponsor: Russian Scientific Medical Society of Therapists (Other)
Responsible Party: Sponsor
Other Study IDs: RNST 01/26
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Cardio-renal-metabolic Syndrome
Keywords: obesity; atherosclerosis; type 2 diabetes mellitus; heart failure
MeSH Terms: conditions — Heart Failure; Obesity; Atherosclerosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study aims to investigate the incidence, associations and prognostic value of CRGM and its components: chronic kidney disease, type 2 diabetes, atherosclerotic cardiovascular diseases, and non-alcoholic fatty liver disease in patients with different phenotypes and severity of clinical manifestations of CHF.

DETAILED DESCRIPTION:
The CARMEN-CHF study is a multicenter, observational, prospective study of the KRGMB in patients with pre-onset CHF or clinically overt CHF.

Patients who meet the study eligibility criteria and consent to participate must provide written informed consent prior to any study-related procedures. By signing the informed consent form, patients grant access to medical information for the purpose of verifying eligibility and collecting information during follow-up.

To ensure a representative sample, it is planned to enroll at least 3,000 patients at study centers across Russia. The proportion of patients included based on pre-onset CHF will be limited to 25% of the entire cohort.

The study's follow-up period is 24 months, during which four visits are planned: two telephone visits at 6 and 18 months, and two in-person visits at 12 and 24 months. If it is not possible to visit a doctor in person, it is permissible to collect information through telephone contacts with the patient or his relative or person caring for the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. A diagnosis that satisfies one of the following criteria:

   * At least one of the following:

LVEF <50%, LV longitudinal systolic strain (GLS) <18%, NT-proBNP >125 pg/mL in sinus rhythm or 365 in AF/AT, E/é >9 at rest by tissue Doppler, Indexed left ventricular volume (ILV) >34 mL/m2 in sinus rhythm or 40 mL/m2 in AF/AT, Tricuspid regurgitation (TR) velocity >2.8 m/s or pulmonary artery systolic pressure (PASP) >35 mmHg. at rest, Left ventricular myocardial mass index (LVMI) >115/95 g/m2 in men/women and relative wall thickness (RWT) >0.42, in the absence of symptoms and/or signs of current or past CHF, which corresponds to "pre-CHF" in accordance with the 2024 clinical guidelines.

or

* LVEF <50% and the presence of symptoms and/or signs of current or past CHF or
* LVEF ≥50% and the presence of symptoms and/or signs of current or past CHF, as well as at least one of the following (A, B, C) criteria:

A. Presence of one of the signs of structural and/or functional heart disorders consistent with the presence of diastolic dysfunction / elevated left ventricular filling pressure:

1. . NT-proBNP level >200 pg/mL in sinus rhythm or >600 pg/mL in AF/AT,
2. . E/é >13 at rest by tissue Doppler,
3. . 13 ≥E/é >9 + left atrial dilation (LAD) >34 ml/m2 in sinus rhythm or >40 ml/m2 in AF/AT,
4. . 13 ≥E/é >9 + TR velocity >2.8 m/s or PASP >35 mmHg at rest,
5. . 13 ≥E/é >9 + presence of left ventricular hypertrophy, defined as LVMI >115 g/m2 in men and >95 g/m2 in women, WCT >0.42, OR B. Presence of 7-9 points on the H2FPEF scale; OR C. Positive diastolic stress test result confirming increased LV filling pressure (E/e'≥15, TR velocity >3.4 m/s) 3. No intravenous therapy with diuretics, nitrates, vasopressors, or inotropes within 24 hours prior to inclusion; 4. Availability of results of all of the following tests, performed no earlier than in the previous 6 months prior to inclusion in the study:

[1] Complete blood count with hemoglobin and platelet levels, [2] Blood chemistry with total bilirubin, ALT, and AST levels, [3] Serum uric acid and creatinine levels, with glomerular filtration rate (eGFR) calculation using the 2021 CKD-EPI formula, [4] Fasting glucose and HbA1c, and, if the diagnosis is uncertain, an oral glucose tolerance test, [5] Ultrasound of the carotid and/or femoral arteries (only in patients with no prior history of atherosclerotic cardiovascular disease), [6] Urine test for CKD markers - at least one of the following: daily albuminuria (mg/day) and/or albumin/creatinine ratio in a single urine portion (mg/g or mg/mmol) and/or daily proteinuria (g/day) and/or protein/creatinine ratio in a single urine portion (mg/g or mg/mmol). -

Exclusion Criteria:

* 1. Current participation in a randomized clinical trial; 2. Confirmed or suspected diagnosis of an alternative or comorbid condition that, in the opinion of the investigator, may explain the patient's symptoms and signs of CHF; 3. History of heart transplantation, combined congenital heart disease, or the presence of a mechanical circulatory support device; 4. Cardiac tamponade; 5. Pregnancy and lactation, planning a pregnancy in the next 24 months; 6. Acute cerebrovascular accident, transient ischemic attack, acute coronary syndrome, or coronary revascularization within less than 30 days prior to or on the day of study inclusion; 7. Acute dysfunction or failure of one or more internal organs within 3 months prior to or on the day of inclusion; 8. Any cardiac surgery performed within 3 months prior to enrollment or planned within the next 6 months, including implantation of intracardiac devices, ablation for cardiac arrhythmias, or correction of valvular pathology; 9. Severe cognitive impairment or other conditions that, in the opinion of the investigator, prevent the patient from understanding the program, providing informed consent, or interfere with participation in the study; 10. Active cancer; 11. Verified cardiac amyloidosis or other infiltrative cardiomyopathy (hemochromatosis, Fabry disease, Gaucher disease); 12. Verified hereditary cardiomyopathy; 13. Heart disease due to reversible causes (e.g., Takotsubo syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with pre-existing or clinically evident CHF at the outpatient stage or in hospital, provided that their condition is stabilized and there has been no intravenous therapy with diuretics, nitrates, vasopressors or inotropes during the previous 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with the presence ofCardio-Kidney-Metabolic (CKM) Syndrome its components and their combinations | From date of enrollment until the date of first documented progression assessed up to 24 months
the proportion of patients with the presence ofCardio-Kidney-Metabolic (CKM) Syndrome its components and their combinations | From date of enrollment until the date of first documented occurrence assessed up to 24 months
  the frequency of occurrence, associations and prognostic value of Cardio-Kidney-Metabolic (CKM) Syndrome and its components (CKD, T2DM, ASCVD and MAFLD) in patients with different phenotypes (hereinafter phenotypes - CHF with reduced, moderately reduced and preserved LVEF) and severity of clinical manifestations of CHF (hereinafter severity of clinical manifestations of CHF - pre-CHF, functional class (FC) I-II and III-IV).

SECONDARY OUTCOMES:
the proportion of patients developing adverse outcomes after 6, 12 and 24 months of follow-up | From date of enrollment until the date of first documented cardiovascular death, • hospitalization due to decompensated CHF, • total number of episodes of CHF worsening, including hospitalizations due to , whichever came first, assessed up to 24 months"
  Determine the proportion of patients developing adverse outcomes after 6, 12, and 24 months of follow-up:
  * cardiovascular death,
  * hospitalization due to decompensated CHF,
  * total number of episodes of CHF worsening, including hospitalizations due to decompensated CHF and outpatient worsening of CHF,
  * death from any cause,
  * death from any cause or hospitalization due to decompensated CHF,
  * hospitalization for any cause,
  * any major cardiovascular event (including cardiovascular death, hospitalization due to decompensated CHF, acute myocardial infarction, unplanned revascularization, new-onset atrial fibrillation (AF), device implantation (cardioverter-defibrillator, pacemaker, cardiac resynchronization therapy device), unplanned cardiac surgery valves, acute cerebrovascular accident, revascularization of the carotid or peripheral arteries);
frequency of transition from pre-CHF to clinically expressed CHF | From the enrollment to the documented clinically expressed CHF assessed up to 24 months
  frequency of transition from pre-CHF to clinically expressed CHF depending on the initial signs of systolic or diastolic dysfunction of the left ventricle, the initial presence of 1, 2, 3 or 4 components of the CRGM, the therapy being administered

CONTACTS AND LOCATIONS:
Overall Officials: Oxana Drapkina, doctor of sciences, Study Chair — National Medical Research Center for Terapy and Preventive Medicine; Anna Chesnikova, doctor of sciences, Study Chair — Rostov-on-Don State Medical Univercity

IPD SHARING:
Plan to Share IPD: Undecided